CLINICAL TRIAL: NCT04586582
Title: The First Affiliated Hospital of Chongqing Medical University.
Brief Title: ST-Segment Resolution as a Marker for Myocardial Scar in ST-Segment Elevation Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Clinical Professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 20180701
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ST-segment resolution <40.15%: ST-segment resolution <40.15%
  Interventions: Diagnostic Test: ST-segment resolution <40.15%
- ST-segment resolution >40.15%: ST-segment resolution >40.15%
  Interventions: Diagnostic Test: ST-segment resolution <40.15%

INTERVENTIONS:
Diagnostic Test: ST-segment resolution <40.15% — Forty-two STEMI patients with single-branch coronary artery stenosis or occlusion were enrolled. ST-segment elevations were measured at emergency admission and at 24 h after PCI. Late gadolinium-enhanced cardiac magnetic resonance imaging (CMR-LGE) was performed 7 days after PCI to evaluate myocardial scars.

SUMMARY:
Clinical studies found that poor ST-segment resolution (STR) in electrocardiogram (ECG) occurred in major adverse cardiovascular events (MACE), arrhythmia and heart failure was significantly higher . In clinical work, in patients have poor ST-segment decline, the investigators found by CMR-LGE the corresponding myocardium become thinner and other signs of myocardial scar.

The investigators aimed to establish whether poor ST-segment resolution in ECG, as well as CMR-LGE, could detect the presence of myocardial scar in early STEMI patients. In order to provide convenient, cheap and widely used test method for patients who cannot tolerate CMR-LGE.

42 STEMI patients with single-branch coronary artery stenosis or occlusion were enrolled. ST-segment elevations were measured on the baseline and 24 hours after PCI. The study population was divided into two groups by late gadolinium enhanced cardiac magnetic resonance (LGE- CMR), with transmural myocardial scar (>75%) or non-transmural myocardial scar (<75%).

ELIGIBILITY:
Inclusion Criteria:

1. Single-branch coronary artery stenosis or occlusion
2. Restoration of coronary perfusion to TIMI flow grade 3 after PCI

Exclusion Criteria:

1. A prior history of the acute coronary syndrome
2. Coronary revascularization
3. Severe chronic kidney disease
4. Intracardiac pacing leads or other implants precluding CMR-LGE
5. Hemodynamic instability
6. Known claustrophobia

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 42 patients.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
ST-segment resolution<40.15% | 1) Emergency admission: ST-segment elevations were measured. 2) 24 hours after PCI: ST-segment elevations were measured. 3) 7 days after PCI: CMR-LGE was performed.
  CMR-LGE was performed to evaluate myocardial scars.
ST-segment resolution>40.15% | 1) Emergency admission: ST-segment elevations were measured. 2) 24 hours after PCI: ST-segment elevations were measured. 3) 7 days after PCI: CMR-LGE was performed.
  CMR-LGE was performed to evaluate myocardial scars.

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, phD., Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The first affiliated hospital of Chongqing medical university, Chongqing, Chongqing Municipality, China